CLINICAL TRIAL: NCT00410176
Title: A Randomized, Controlled, Unblinded, Clinical Trial of the Acceptability and Efficacy of Non-Pharmaceutical Methods in Preventing Spread of Influenza Within the Family
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Israel (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4335CTIL
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Sanitation

INTERVENTIONS:
Behavioral: sanitation and personal hygiene

SUMMARY:
The proposed study will evaluate whether the use of non-pharmaceutical methods, such as surgical masks, isolation of patients and personal hygiene, are acceptable and effective in preventing the spread of influenza within the family.This will be achieved by conducting a randomized, controlled, unblinded, clinical trial. Family members of an index case with influenza like illness, will be randomly allocated to two groups. In the intervention group, family members will receive comprehensive guidance about sanitation and hygiene, as well as surgical masks to wear whenever in close contact (3 feet / 1 meter) with the index case. In addition, they will be asked to isolate the index case as much as possible. In the control group, family members will receive only standard guidance about sanitation and hygiene relevant for reducing the transmission of influenza. The primary end-point of the study will be secondary infection of influenza of at least one of the family members in order to asses the efficacy of the interventions. In addition, the compliance to those interventions will be evaluated.

The study hypothesis is that use of non-pharmaceutical methods will be acceptable and will reduce the secondary infection rate among them by 50%.

ELIGIBILITY:
Inclusion Criteria:

* Family members of an index case with influenza-like illness (ILI) during the first two days of his illness.
* No limitations will be given regarding the number of family members.

Exclusion Criteria:

* Presence of another household member with ILI during the previous two weeks.

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2007-01

PRIMARY OUTCOMES:
secondary infection of influenza within the family

SECONDARY OUTCOMES:
compliance of non-pharmaceutical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Manfred S Green, PhD, M.D, Principal Investigator — ICDC